CLINICAL TRIAL: NCT05851963
Title: Comparison of the Effectiveness of Manual and Electric Toothbrushes in Daily Practice in Patients with Fixed Orthodontic Appliances
Brief Title: Toothbrushes in Daily Practice in Patients with Fixed Orthodontic Appliances
Acronym: ORTHO-IOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Collaborators: University of Nancy (Other)
Responsible Party: Principal Investigator, Carrouel Florence, Associate professor, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ORTHO-IOP
Record Dates: First submitted 2023-03-30; First posted 2023-05-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-08

CONDITIONS: Dental Malposition
Keywords: toothbrush; oral prophylaxis; adolescents; orthodontic appliances

STUDY DESIGN:
Intervention Model Description: Parallel Assignment This trial is designed as an four-arm parallel cluster randomized controlled trial and an allocation ratio of 1:1:1:1
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group using sonic toothbrush (Experimental): Patients will be asked to use a sonic toothbrush for 24 months
  Interventions: Device: Sonicare Diamond Clean 9000
- Group using hydrosonic toothbrush (Experimental): Patients will be asked to use a hydrosonic toothbrush for 24 months
  Interventions: Device: HydroSonic Pro
- Group using manual toothbrush (Placebo Comparator): Patients will be asked to use a manual toothbrush for 24 months
  Interventions: Device: Oral-B 123
- Group using manual toothbrush with 5460 strands (Experimental): Patients will be asked to use a manual toothbrush with 5460 strands for 24 months
  Interventions: Device: Curaprox CS 5460

INTERVENTIONS:
Device: Sonicare Diamond Clean 9000 — Brush teeth with the electric toothbrush 1 daily during the orthodontic treatment
  Arms: Group using sonic toothbrush
Device: HydroSonic Pro — Brush teeth with the electric toothbrush 2 daily during the orthodontic treatment
  Arms: Group using hydrosonic toothbrush
Device: Oral-B 123 — Brush teeth with the electric toothbrush 2 daily during the orthodontic treatment
  Arms: Group using manual toothbrush
Device: Curaprox CS 5460 — Brush teeth with the electric toothbrush 2 daily during the orthodontic treatment
  Arms: Group using manual toothbrush with 5460 strands

SUMMARY:
Because of the difficulties of disorganizing the dental biofilm in these adolescents with fixed orthodontic treatment, electric toothbrushes have been proposed as an alternative to manual toothbrushes. Electric toothbrushes, available in a wide range of price points, have been developed with the goal of replicating the complex motions required by the manual toothbrush and making plaque removal more efficient. However, the overall effect size is limited, and the clinical relevance is not yet clear. Applied to orthodontics, specialized manual toothbrushes have also recently been developed. Few recent clinical trials have been conducted in patients with orthodontic appliances.

Thus, the question of whether and which type of manual or electric toothbrushes may be beneficial for patients with orthodontic appliances is still unresolved. Given the variety of toothbrushes available on the market, there is a need for sound clinical research to evaluate their effectiveness to guide professional recommendations. This work will provide a significant advance in the knowledge of the potential of the latest generation of electric toothbrushes on gingival inflammation, potentially reducing the risk of caries and gingival lesions.

ELIGIBILITY:
Inclusion Criteria:

* Children to be treated with fixed upper and lower braces
* 11 to 15 years of age at the start of treatment
* One parent/legal guardian agrees to the terms and conditions of the study and signs the informed consent form
* The adolescent agrees to the terms and conditions of the study and signs the informed consent form

Exclusion Criteria:

* Less than 20 permanent teeth with braces or brackets
* Presence of untreated cavities
* Bleeding greater than 10% on probing
* Presence of a gingival pocket larger than 5 mm
* Presence of fixed prosthetic restorations
* Presence of any enamel development defect
* Presence of dental anomalies or direct/indirect labial restorations on teeth
* Patients requiring orthognathic surgeries
* Presence of systemic diseases (diabetes, hepatic, renal, hematologic, cardiovascular)
* Use of medications that may affect gingival health (such as calcium channel blockers, ciclosporin and anticoagulants)
* Use of antibiotics and anti-inflammatory drugs for any purpose over a long period of time.
* Having a smoking habit
* Having a physical or mental problem that affects manual dexterity
* Being unable to answer questions or being uncooperative

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of gingival bleeding from baseline during orthodontic treatment | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  Change of gingival inflammation in patients with fixed orthodontic appliances using manual or electric toothbrushes in daily practice

SECONDARY OUTCOMES:
Acceptability | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  Questionnaire to assess the acceptability of oral hygiene products by patients
Effect on gingival inflammation | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  gingival index
Effect on gingival bleeding | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  Bleeding on Probing
Effect on dental plaque | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  plaque index
Effect on gingival tissue | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  micro-osteoperforation
Effect on gingival attachment | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  clinical attachment loss
Enamel lesions | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  Assess the incidence of initial enamel lesions
Dentinal hypersensitivity | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  Assess the incidence of dentinal hypersensitivity
Salivary acidity | T1 (1 month), T2 (+ 3 months) and T3 (+ 6 months), T4 (+ 12 months), T5 (+ 15 months) T6 (+ 18 months) and T7 (+ 24 months)
  Measure of pH

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de soin dentaire, Nancy, France

IPD SHARING:
Plan to Share IPD: No